CLINICAL TRIAL: NCT06657274
Title: EARLY-COGN^3 - Smart Digital Solutions for EARLY Treatment of COGnitive Disability: a Neuropsychological, Neurophysiological and Neurobiological Perspective in Chronic Neurological Diseases - PNRR-MCNT2-2023-12377069
Acronym: EARLY-COGN^3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: European Union - NextGenerationEU - PNRR M6C2 - Mission M6 - Component C2 - Investment 2.1 - Valorizzazione e potenziamento della ricerca biomedica del SSN (Unknown); IRCCS Fondazione Don Carlo Gnocchi, Milano (Unknown); National Research Council (CNR) - Institute for Biomedical Research and Innovation (IRIB), Messina (Unknown); IRCCS Centro Neurolesi Bonino Pulejo, Messina (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EARLY-COGN^3 - PNRR-MCNT2-2023
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment (MCI); Subjective Cognitive Complaints (SCCs); Parkinson Disease
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tele@cognitive treatment (Experimental): The tele@cognitive treatment group will receive a total of 5 weeks (3 sessions/week, 45 minutes/session) of home-based cognitive rehabilitation activities delivered through a digital telerehabilitation platform.
  Interventions: Device: RICORDO-DTx
- Active Control Group (ACG) (Active Comparator): The Active Control Group (ACG), will receive at-home unstructured cognitive stimulation for 5 weeks (3 sessions/week, 45 minutes/session).
  Interventions: Behavioral: Home-based unstructured cognitive stimulation

INTERVENTIONS:
Device: RICORDO-DTx — Tele@cognitive treatment group will receive a total of 5 weeks (3 sessions/week, 45 minutes/session) of home-based cognitive rehabilitation activities with an innovative digital solution for remote rehabilitation of cognitive difficulties according to digital therapeutics delivery model. Subjects assigned to the tele@cognitive group can access the app RICORDO-DTx through a tablet showing the prescribed rehabilitation activities to be performed.
  Each cognitive exercise is structured into five levels of difficulty that adaptively increase (algorithm on both subject's performance and perceived difficulty). All data about patient progress and adherence will be collected with this digital solution and will be available to evaluate and monitor the results of rehabilitation.
  Arms: tele@cognitive treatment
Behavioral: Home-based unstructured cognitive stimulation — Subjects assigned to the home-based unstructured cognitive stimulation will be requested to work on detailed activities for the same duration of the tele@cognitive intervention (3 sessions/week, 45 minutes/session). They will receive, from the therapist, an instructions booklet and a participant diary.
  Arms: Active Control Group (ACG)

SUMMARY:
The increase in life expectancy in recent decades has led to a large number of people living into old age and an increased risk of developing Chronic Neurological Diseases (CNDs) such as neurodegenerative diseases. A higher cumulative risk of dementia has been largely demonstrated in Mild Cognitive Impairment (MCI) and Subjective Cognitive Complaints (SCCs) subjects and in Parkinson's Disease (PD) patients, as compared to the general population. These disorders result in an impairment of the individual's abilities to perform daily tasks. As their disease progresses, patients become dependent on medical services and on family support. Given the limited effectiveness of pharmacological treatments, non-pharmacological interventions to prevent and treat cognitive deficits and the associated difficulties with activities of daily living in neurodegenerative disease patients have gained attention in recent years and, among these, cognitive training offers a potential approach for dementia prevention and improvement of cognitive function. A critical aspect of cognitive training programs is that the most promising interventions have involved intensive in-person sessions that are unlikely to be cost-effective or feasible for large-scale implementation. Within the framework of non-pharmacological interventions, the use of technology to assist the person at risk and/or with mild dementia at home and to extend rehabilitation services in the treatment of dementia has gradually gained importance. Telerehabilitation technologies allow to provide services remotely in patients' homes, allowing access to health care to patients living in rural settings or with mobility difficulties. In addition, the telerehabilitation modality offers the advantage of providing rehabilitation within the natural environment of the patient's home, making the treatment more realistic and possibly more generalizable to the person's daily life. The present project proposes to test a home-based asynchronous cognitive telerehabilitation program aimed at enhancing the continuum of care for MCI, SCCs and PD, using technology. The proposed study is a single blind randomized controlled trial (RCT) involving subjects with CNDs randomly assigned to one out of two intervention groups: i) the tele@cognitive group, who will receive at-home cognitive telerehabilitation (tele@cognitive treatment); ii) the Active Control Group (ACG), who will receive at-home unstructured cognitive stimulation. The aim of the project will be threefold: [1] to test the short-term and long-term efficacy of tele@cognitive protocol as compared to an unstructured cognitive at-home rehabilitation in the treatment of a cohort of patients with CNDs; [2] to explore the changes induced by tele@cognitive intervention on biomolecular and neurophysiological markers; [3] to explore potential cognitive, neurobiological and neurophysiological predictors of response to tele@cognitive treatment.

DETAILED DESCRIPTION:
60 subjects with MCI, SCC, PD will be recruited from IRCCS Istituto Centro San Giovanni di Dio, Fatebenefratelli, Brescia, Fondazione Don Carlo Gnocchi - ONLUS, Milan and IRCCS Centro Neurolesi Bonino Pulejo, Messina.

Patients will include both male and female subjects affected by CND: PD (Hoehn & Yahr<3), MCI (with CDR scale≤0.5, MMSE ≥24) and SCC (Subjective Cognitive Complaints).

All patients will undergo treatment sessions of 45 minutes, 3 days a week for 5 weeks:

* 30 subjects will be assigned to the tele@cognitive group that will receive home-based cognitive telerehabilitation activities with an innovative digital solution for remote rehabilitation of cognitive difficulties according to the digital therapy delivery model;
* 30 subjects will be assigned to the Active Control Group (ACG) that will receive home-based unstructured cognitive stimulation.

The two groups will be matched for sex, age, education and performance in the MoCA test.

All study participants will be administered a multidimensional assessment by an experienced neuropsychologist at baseline (T0), at post-treatment assessment (T1, 5 weeks from T0) and at 3-month follow-up (T2). In addition, participation in the research involves blood sampling and application of Transcranial Magnetic Stimulation (TMS) before (T0) and after (T1) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD (Hoehn & Yahr<3); MCI (with CDR scale≤0.5, MMSE ≥24), and SCC (Subjective Cognitive Complaints);
* Montreal Cognitive Assessment (MoCA) corrected score ≥17.36
* Education ≥ 5 years
* Age eligible for the study: 18≤age≤85
* Native Italian speakers
* Absence of marked hearing/visual impairment
* All of the subjects will have normal or corrected-to-normal vision.
* Agreement to participate by signing the informed consent form
* Availability of a caregiver/study partner able to support the participant
* No rehabilitation program in place at the time of enrolment or in the last 3 months before enrolment
* Stable drug treatment (last 3 months), if any

Exclusion Criteria:

* Presence of any medical or psychiatric illness that could interfere with completing assessments;
* Presence of any medical condition representing a contraindication to TMS.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in global cognition as assessed by Montreal Cognitive Assessment (MoCA) | Baseline up to 5 weeks and 3 months
  Montreal Cognitive Assessment (MoCA) is a screening test for global cognitive functioning. It includes tasks involving several cognitive domains: visuospatial, executive function, naming, selective and sustained attention, language, abstraction, memory and orientation (score range min= 0, max= 30, higher score=better outcome).
Change in long-term episodic verbal memory as assessed by Free and Cued Selective Reminding Test (FCSRT) | Baseline up to 5 weeks and 3 months
  Free and Cued Selective Reminding Test (FCSRT) is a measure of long-term episodic verbal memory. It provides five scores: Immediate Free Recall (IFR, spontaneous recall across three trials; score range min= 0, max= 36), Immediate Total Recall (ITR, total recall across three trials; score range min= 0, max= 36), Delayed Free Recall (DFR, score range min= 0, max= 12), Delayed Total Recall (DTR, score range min= 0, max= 12). Higher scores indicate better performance. Finally, the Index of Sensitivity to Cueing (ISC, score range min= 0, max= 1) reflects the difference between the number of items recalled spontaneously and the number of items recalled with the help of cues. A higher ISC indicates a greater sensitivity to cues.

SECONDARY OUTCOMES:
Change in measure of quality of life as assessed by EQ-5D-5L | Baseline up to 5 weeks and 3 months
  EQ-5D-5L is a measure of health status consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has three response levels (no problems, some problems, unable to/extreme problems). In addition, the questionnaire includes a visual analog scale that records the patient's perception of his or her overall health (score range: min= 0, max= 100, higher score=better outcome).
Change in measure of non-motor experiences of daily living as assessed by MDS-UPDRS scale, part I | Baseline up to 5 weeks and 3 months
  MDS-UPDRS scale, part I (only for PD patients) is a measure of non-motor experiences of daily living consisting of a total of 13 questions (score range min= 0, max= 52, higher score= worse outcome).
Change in measure of motor abilities as assessed by MDS-UPDRS scale, part III | Baseline up to 5 weeks and 3 months
  MDS-UPDRS scale, part III (only for PD patients) is a measure of motor abilities consisting of a total of 18 questions with 33 individual items. Each item has a 0-4 rating, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe (score range: min= 0, max= 132, higher score=worse outcome).
Change in depressive symptoms as assessed by Hamilton Depression Rating Scale (HDRS) | Baseline up to 5 weeks and 3 months
  Hamilton Depression Rating Scale (HDRS) is a measure of severity of depressive symptoms consisting of a total of 21 items (score range min= 0, max= 64, higher score=worse outcome).
Change in anxiety symptoms as assessed by State-Trait Anxiety Inventory (STAI-Y) | Baseline up to 5 weeks and 3 months
  The STAI-Y consisting of two 20-item scales providing separate measures of state and trait anxiety (S-Anxiety and T-Anxiety). Each scale has a score range from a minimum of 20 to a maximum of 80 and a higher score on the scale indicates a worse outcome.
Change in behavior and personality as assessed by Neuropsychiatric Inventory (NPI) | Baseline up to 5 weeks and 3 months
  Neuropsychiatric Inventory (NPI) is used for assessing various neuropsychiatric symptoms. The inventory consists of 12 core domains, each reflecting specific neuropsychiatric symptoms. Each symptom is rated for both frequency and severity. (score range min= 0, max= 144, higher score=worse outcome).
Change in memory complaints as assessed by Everyday Memory Questionnaire (EMQ) | Baseline up to 5 weeks and 3 months
  Everyday Memory Questionnaire (EMQ) is a 20-items questionnaire that evaluate the frequency and impact of memory problems in daily life (score range min= 20, max= 180, higher score=worse outcome).
Change in non-verbal abstract reasoning as assessed by Raven's Coloured Progressive Matrices | Baseline up to 5 weeks and 3 months
  Raven's Coloured Progressive Matrices is a measure of non-verbal abstract reasoning (score range min= 0, max= 36, higher score=better outcome).
Change in measure of attentional abilities as assessed by Trial Making Test (TMT) | Baseline up to 5 weeks and 3 months
  Trial Making Test (TMT, part-A and part-B) is a measure of attentional abilities, visuo-conceptual and visual-motor tracking. TMT-Part A involves visual scanning, number recognition, number sequencing and motor speed. TMT-Part B assesses mental flexibility in managing more than one stimulus at a time and in shifting the course of an ongoing activity. High execution times indicate poor performance (score range: min= n/a, max= no limits).
Change in measure of executive abilities as assessed by Stroop Test | Baseline up to 5 weeks and 3 months
  Stroop Test is a measure of executive abilities, including visual attention, selective attention, cognitive flexibility and inhibitory control of behavior. Two scores are calculated considering the number of errors and the time taken to complete all parts. High execution times and high numbers of errors indicate poor performance.
Change in measure of constructional praxia as assessed by Rey-Osterrieth Complex Figure-Copy | Baseline up to 5 weeks and 3 months
  Rey-Osterrieth Complex Figure-Copy is a measure of constructional praxia (score range min= 0, max= 36, higher score=better outcome).
Change in measure of fluency abilities as assessed by Verbal Fluency (semantic and phonemic) | Baseline up to 5 weeks and 3 months
  Verbal Fluency (semantic and phonemic) is a measure of verbal and semantic fluency abilities, executive functions abilities, lexical store size, lexicon access, and lexical organization (score range min= 0, max= no limits, higher score=better outcome).
Change in measure of nonverbal long-term memory as assessed by Rey-Osterrieth Complex Figure-Recall | Baseline up to 5 weeks and 3 months
  Rey-Osterrieth Complex Figure-Recall is a measure of nonverbal long-term memory (score range min= 0, max= 36, higher score=better outcome).
Change in NFL and Tau | Baseline up to 5 weeks
  Neurofilament light chain (NFL) and Tau levels
Change in Aß1-40, Aß1-42, p-tau-181; p-tau-231, alpha-synuclein | Baseline up to 5 weeks
  Aß1-40, Aß1-42, p-tau-181; p-tau-231, alpha-synuclein levels
Change in GFAP, chemokines and sTREM2 | Baseline up to 5 weeks
  Glial Fibrillary Acidic Protein (GFAP), chemokines and sTREM2 levels
Change in Neurogranin and BDNF | Baseline up to 5 week
  Neurogranin and Brain-Derived Neurotrophic Factor (BDNF) levels
Change in plasma EVs | Baseline up to 5 weeks
  Size and the concentration of plasma Extracellular Vescicles (EVs)
Change in rMT | Baseline up to 5 weeks
  TMS resting Motor Threshold (rMT)
Change in MEPs | Baseline up to 5 weeks
  TMS Motor Evoked Potentials (MEPs)
Change in SICI | Baseline up to 5 weeks
  TMS Short-interval intracortical inhibition (SICI)
Change in SAI | Baseline up to 5 weeks
  TMS Short-latency afferent inhibition (SAI)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, IT
  - IRCCS Centro Neurolesi Bonino Pulejo, Messina, IT
  - Fondazione Don Carlo Gnocchi - ONLUS, Milan, Milan, IT

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cotelli M, Baglio F, Gobbi E, Campana E, Pagnoni I, Cannarella G, Del Torto A, Rossetto F, Comanducci A, Tartarisco G, Calabro RS, Campisi S, Maione R, Saraceno C, Dognini E, Bellini S, Bortoletto M, Binetti G, Ghidoni R, Manenti R. Smart Digital Solutions for EARLY Treatment of COGNitive Disability (EARLY-COGN;3): A Study Protocol. Brain Sci. 2025 Feb 24;15(3):239. doi: 10.3390/brainsci15030239. PMID 40149761